CLINICAL TRIAL: NCT01380015
Title: Human Clinical Trial to Investigate the Effects of High Rosmarinic Acid Spearmint Tea on Markers of Pain, Physical Function and Disease Activity in Osteoarthritis of the Knee
Brief Title: Efficacy of Spearmint Tea in Relieving Osteoarthritis of the Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Ontario Ministry of Agriculture, Food and Rural Affairs (Other Government)
Responsible Party: Principal Investigator, Amanda Wright, Ph.D., Director, HNRU, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 11JA040
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; spearmint; rosmarinic acid
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Control (Placebo Comparator): Participants will consume two cups of commercial spearmint tea per day (300 mL in the morning and 300 mL in the evening, providing a total of approximately 20 mg of rosmarinic acid per day) for a total of 4 months.
  Interventions: Other: Commercially spearmint tea
- Experimental (Experimental): Participants will consume two cups of a high rosmarinic acid spearmint tea per day (300 mL in the morning and 300 mL in the evening, providing a total of approximately 300 mg of rosmarinic acid per day) for a total of 4 months.
  Interventions: Other: High Rosmarinic Acid Spearmint Tea

INTERVENTIONS:
Other: Commercially spearmint tea — Commercially available, non-selectively bred spearmint tea.
  Arms: Placebo Control
Other: High Rosmarinic Acid Spearmint Tea — The investigational product will be a high rosmarinic acid spearmint tea (700B) developed by the Department of Plant Agriculture, University of Guelph. Clone 700B has been selectively bred to contain a rosmarinic acid content 15-20 times greater than that of typical mint.
  Arms: Experimental

SUMMARY:
The purpose of this study is to investigate the benefits of daily consumption of a high rosmarinic acid spearmint tea, developed by the University of Guelph, on measures of pain, physical function and disease activity in osteoarthritis of the knee.

The investigators hypothesize that a spearmint tea high in rosmarinic acid is efficacious in mitigating the symptoms of osteoarthritis of the knee through its actions in reducing cartilage degradation, oxidative stress and inflammation.

DETAILED DESCRIPTION:
Healthy adults with a clinical diagnosis of osteoarthritis of the knee will be recruited and will undergo a brief phone screening interview, followed by a detailed in-person screening process, to determine study eligibility.

Eligible participants will be matched according to sex, baseline pain according to the Western Ontario and McMaster Universities Arthritis Index (WOMAC) score, and duration of osteoarthritis. Participants will then be randomly assigned to receive either the investigative high rosmarinic acid spearmint tea or a comparable placebo mint tea.

During the 4-month treatment period, participants will consume two cups (300 mL in the morning and 300 mL in the evening) of either the high rosmarinic acid spearmint tea (approximately 300 mg rosmarinic acid per day) or the commercial spearmint tea (approximately 20 mg of rosmarinic acid per day) daily.

Data collection will occur at baseline (week 0), mid-treatment (week 8), post-treatment (week 16), and follow-up (week 20). Outcome measures include WOMAC and SF-36 scores, physical function (6-minute walk, stair climb task), inflammatory markers (serum C-reactive protein), and self-reported changes in pain medication use. In a sub-set of consenting participants deemed eligible by the study physician, a synovial fluid sample will be drawn from the knee for the analyses of cartilage degradation biomarkers (GAG, COMP, PGE2, NO) at baseline (week 0) and post-treatment (week 16).

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years or older
* Have been diagnosed by a health care professional with osteoarthritis of the knee
* Demonstrates a WOMAC pain score greater then 125 at time of study screening

Exclusion Criteria:

* Has any other systemic or rheumatic arthritis
* Has completed or is planning to undergo knee replacement surgery
* Has had a chemical, radiologic, or surgical synovectomy in any large joint within the previous 3 months
* Has any concomitant inflammatory processes such as infectious or rheumatic disease
* Has any gastrointestinal ulcers
* Has any clinically significant, uncontrolled cardiovascular, hepatic, renal, or any other medical condition that may interfere with the study
* Has any serious medication conditions such as recent (within the previous 6 months) heart attack, stroke, cancer and/or diabetes
* Has a recent history (within the previous 6 months) of a clinically significant psychiatric disorder other than mild depression
* Has a known allergy or hypersensitivity to mint or any other food allergies
* Smokes, drinks alcohol (>14 drinks per week) or participates in recreational drug use
* Has participated in a clinical trial involving an investigational or marketed drug within the previous 6 months
* Women who are pregnant or plan to become pregnant during the study period, women who have recently (within the previous 6 months) given birth, women who are currently lactating or have only recently (within the previous 6 months) stopped lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Self-reported ratings of pain and physical function | Four months
  Data collection of self-reported ratings of pain and physical function (WOMAC), self-reported ratings of overall physical and mental health (SF-36), and self-reported changes in the use of concomitant pain and inflammation medications (study diary) will occur at baseline (week 0), mid-treatment (week 8), post-treatment (week 16), and follow-up (week 20).
Use of concomitant pain/inflammatory medications for the management of osteoarthritis symptoms | Four months

SECONDARY OUTCOMES:
Performance-based measures of physical function | Four months
  Data for performance-based assessment of physical function (6-minute walk, stair climb task) will be collected at baseline (week 0), mid-treatment (week 8), post-treatment (week 16), and follow-up (week 20).
Change in synovial fluid biomarkers of cartilage degradation | Four months
  In a sub-set of participants, a synovial fluid sample will be drawn (i.e. arthocentesis) for the analyses of cartilage degradation biomarkers (GAG, COMP, PGE2, NO) at baseline (week 0) and post-treatment (week 16).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda J Wright, Ph.D., Principal Investigator — Human Nutraceutical Research Unit; Alison M Duncan, Ph.D., R.D., Principal Investigator — Human Nutraceutical Research Unit
Locations (2):
- Canada (2):
  - University of Guelph, Guelph, Ontario
  - Human Nutraceutical Research Unit, University of Guelph, Guelph, Ontario

REFERENCES:
- [Derived] Connelly AE, Tucker AJ, Tulk H, Catapang M, Chapman L, Sheikh N, Yurchenko S, Fletcher R, Kott LS, Duncan AM, Wright AJ. High-rosmarinic acid spearmint tea in the management of knee osteoarthritis symptoms. J Med Food. 2014 Dec;17(12):1361-7. doi: 10.1089/jmf.2013.0189. PMID 25058311